CLINICAL TRIAL: NCT00316901
Title: PET/CT Evaluation of Subjects Treated on Surgery Branch Adoptive Cell Therapy Protocols
Brief Title: Positron Emission Tomography and CT Scan in Predicting Response in Patients With Metastatic Melanoma or Kidney Cancer Who Are Undergoing Cellular Adoptive Immunotherapy on a Surgery Branch Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 060099; 06-C-0099; NCI-P6831; CDR0000470868
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage IV renal cell cancer; stage IV melanoma; recurrent melanoma; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

INTERVENTIONS:
Procedure: computed tomography
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography and computed tomography scan (done before and after cellular adoptive immunotherapy), may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II trial is studying how well positron emission tomography and computed tomography scan predicts response in patients with metastatic melanoma or kidney cancer who are undergoing cellular adoptive immunotherapy on a Surgery Branch clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Measure changes in metabolic activity at visceral sites during the acute treatment phase of adoptive cell transfer (ACT) using positron emission tomography (PET)/CT fusion imaging in patients with metastatic melanoma or renal cell cancer.
* Measure changes in metabolic activity at metastatic sites during the acute treatment phase of ACT using PET/CT fusion imaging.
* Compare the changes in metabolic activity at visceral and metastatic sites in patients treated with intravenous vs intra-arterial tumor-infiltrating lymphocyte infusions.

Secondary

* Correlate response of individual metastases with these metabolic alterations.

OUTLINE: This is a pilot study. Patients are stratified according to treatment (intravenous [IV] tumor-infiltrating lymphocytes [TIL] after a nonmyeloablative preparative regimen vs intra-arterial [IA] TIL after a nonmyeloablative preparative regimen vs IV TIL after a myeloablative preparative regimen with chemotherapy and total-body irradiation).

Patients undergo positron emission tomography with fludeoxyglucose F 18 (FDG-PET)/CT fusion imaging at baseline (before starting TIL infusion), once between days 1-4 after TIL infusion, and once between days 5-8 after TIL infusion.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Melanoma
  * Renal cell cancer
* Metastatic disease
* Measurable disease by CT scan or MRI
* Enrolled in a Surgery Branch protocol utilizing 1 of the following variations of adoptive cell transfer of tumor-infiltrating lymphocytes (TIL):

  * Intravenous (IV) TIL after a nonmyeloablative preparative regimen (e.g., NCI-99-C-0158)
  * Intra-arterial (IA) TIL after a nonmyeloablative preparative regimen (e.g., NCI-99-C-0158)
  * IV TIL after a myeloablative preparative regimen with chemotherapy and total-body irradiation (e.g., NCI-04-C-0288)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No history of or treatment for diabetes mellitus
* No hypersensitivity or allergy to fludeoxyglucose F 18
* Weight ≤ 350 lbs (136 kg)
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No treatment with both IV and IA TIL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Metabolic activity at visceral sites
Metabolic activity at metastatic sites
Differences in metabolic activity at visceral and metastatic sites in patients treated with intravenous and intraarterial cell infusions

SECONDARY OUTCOMES:
Response of individual metastases in comparison with metabolic alterations

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Royal, MD, FACS, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States